CLINICAL TRIAL: NCT06254378
Title: Evaluation of the Efficacy of Allograft Versus Tenting Technique in Open Sinus Lifting With Immediate Implant Placement A Randomized Clinical Trial
Brief Title: Evaluation of the Efficacy of Allograft Versus Tenting Technique in Open Sinus Lifting With Immediate Implant Placement
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Amira Raafat Ahmed Elshikh, Dentist, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Sinus lifting
Record Dates: First submitted 2024-01-25; First posted 2024-02-12 (Actual); Last update posted 2024-02-12 (Actual); Status verified 2024-01

CONDITIONS: Sinus; Dental; Implant Complication; Surgery-Complications
MeSH Terms: conditions — Fistula | interventions — Transplantation, Homologous; Transplantation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sinus lifting without graft (control ) (Active Comparator): Patients will receive sinus lifting with immediate implant placement without graft placement.
  Interventions: Other: Sinus lifting without graft
- Sinus lifting with graft (intervention) (Experimental): Patients will receive sinus lifting with immediate implant and allograft placement.
  Interventions: Procedure: Sinus lifting with allograft

INTERVENTIONS:
Procedure: Sinus lifting with allograft — Participants will receive sinus lifting and allograft with immediate implant in premolar-molar area.
  Arms: Sinus lifting with graft (intervention)
Other: Sinus lifting without graft — Participants will receive sinus lifting with immediate implant in premolar-molar area without graft
  Other Names: Tenting technique
  Arms: Sinus lifting without graft (control )

SUMMARY:
Implant placement in deficient posterior maxilla is a challenging clinical situation that necessitates appropriate treatment options to restore this area.

-Aim of the study: To compare allograft vs tenting technique in terms of implant stability and bone height.

DETAILED DESCRIPTION:
Rationale for carrying out the trial:

The research population will be divided into two groups. Group1 will be treated by allograft with immediate implant technique, Group2 will be treated by tenting technique with immediate implant technique. Allograft has been effective in augmenting bone growth and has been proven to be a vital asset in sinus lifting.

ELIGIBILITY:
Inclusion Criteria:

1. Patient with missing upper pre molar , molar teeth
2. Patients in need of bone grafting of the maxillary sinus to house an implant.
3. Patients with residual alveolar crest of at least 3-4mm in height and 5mm in width distal to the canine as measured on CBCT scan
4. Patients with adequate inter-arch space

Exclusion Criteria:

1. Patients suffering from any sinus pathosis.
2. Patients who are heavy smokers (>10 cigarettes/day).
3. Patient under psychiatric therapy or unrealistic expectations
4. Patients of systemic conditions that may interfere with carrying out the surgical procedure.
5. Lack of opposite occluding dentition/prosthesis in the area intended for implant placement
6. Severe bruxism or clenching
7. Poor oral hygiene (full mouth bleeding on probing and full mouth plaque index >25%)

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-03-01 (Estimated); Primary Completion 2024-09-30 (Estimated); Study Completion 2024-10-30 (Estimated)

PRIMARY OUTCOMES:
Implant stability | During the implant placement procedure and after 6 months
  implant stability quotient(ISQ) is the evaluation unit set to determine the correct isq<60:low stability isq 60-65 : medium stability isq >70: high stability stability of the implant, this module by means of a resonance frequency analysis (rfa) applied to the bone manages to measure stability on an isq scale from 1 to 100 (khz):

SECONDARY OUTCOMES:
Bone hight | Before surgery and after 6 months
  Newly formed bone length will be measured on cone beam ct by millimeter

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fouad W, Osman A, Atef M, Hakam M. Guided maxillary sinus floor elevation using deproteinized bovine bone versus graftless Schneiderian membrane elevation with simultaneous implant placement: Randomized clinical trial. Clin Implant Dent Relat Res. 2018 Jun;20(3):424-433. doi: 10.1111/cid.12601. Epub 2018 Mar 25. PMID 29575547
- [Result] Karagah A, Tabrizi R, Mohammadhosseinzade P, Mirzadeh M, Tofangchiha M, Lajolo C, Patini R. Effect of Sinus Floor Augmentation with Platelet-Rich Fibrin Versus Allogeneic Bone Graft on Stability of One-Stage Dental Implants: A Split-Mouth Randomized Clinical Trial. Int J Environ Res Public Health. 2022 Aug 4;19(15):9569. doi: 10.3390/ijerph19159569. PMID 35954926